CLINICAL TRIAL: NCT01028534
Title: Comparison of the Effects of Different Antihypertensive Drugs in Patients With Hypertension and Obstructive Sleep Apnea
Brief Title: Effects of Antihypertensive Drugs in Patients With Hypertension and Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Toru Oga, Respiratory Care and Sleep Control Medicine, Kyoto University, Graduate School of Medicine, Kyoto University, Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C359kyoto
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Obstructive Sleep Apnea; Hypertension
Keywords: Continuous positive pressure ventilation; Blood pressure; Oxygen desaturation index; Endothelial dysfunction; Patient reported measurement
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension | interventions — olmesartan; azelnidipine; Angiotensin Receptor Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ARB plus increased ARB (Active Comparator): angiotensin II receptor blockers for the first 3 months and increasing dose of angiotensin II receptor blockers for the next 3 months
  Interventions: Drug: Olmesartan and Azelnidipine
- ARB plus CCB (Active Comparator): angiotensin II receptor blockers for the first 3 months and adding calcium channel blockers for the next 3 months
  Interventions: Drug: Olmesartan and Azelnidipine
- CCB plus ARB (Active Comparator): calcium channel blockers for the first 3 months and adding angiotensin II receptor blockers for the next 3 months
  Interventions: Drug: Olmesartan and Azelnidipine

INTERVENTIONS:
Drug: Olmesartan and Azelnidipine — 1. Olmesartan 20mg per day for 3 months and, if hypertension is not controlled, increase Olmesartan to 40mg per day for the next 3 months
  2. Olmesartan 20mg per day for 3 months and, if hypertension is not controlled, add Azelnidipine 16mg per day for the next 3 months
  3. Azelnidipine 16mg per day for 3 months, and, if hypertension is not controlled, add Olmesartan 20mg per day for the next 3 months
  Other Names: Olmesartan (angiotensin II receptor blockers: ARB); Azelnidipine (long-acting calcium channel blockers: CCB)

SUMMARY:
The aim of the present study is to compare the effects of different types of antihypertensive drugs (angiotensin II receptor blockers and long-acting calcium channel blockers) in patients with hypertension and obstructive sleep apnea who are not controlled well with their hypertension after continuous positive airway pressure therapy.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) and hypertension have a significant interrelationship, and both disorders are well known risk factors for cardiovascular diseases (CVD). Treating them appropriately may improve the prognosis of the patients. Presently, continuous positive airway pressure (CPAP) therapy is the first-line therapy for OSA, and angiotensin II receptor blockers and long-acting calcium channel blockers for hypertension in Japan. Therefore, in the present study, we wanted to compare the effects of these different types of antihypertensive drugs on the control of blood pressure in patients with OSA whose hypertension is not controlled well after CPAP therapy.

ELIGIBILITY:
Inclusion Criteria:

* Apnea and hypopnea index of more than 20 /hr, and treated with CPAP
* Uncontrolled hypertension (defined as systolic blood pressure of more than 130 mmHg or diastolic blood pressure of more than 80 mmHg

Exclusion Criteria:

* Cerebrovascular diseases, myocardial infarction, angina pectoris or heart failure within 6 months
* Uncontrolled arrhythmia
* Severe hepatic or renal disorders
* Having poor prognosis disorders such as malignant disorders

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Six months

SECONDARY OUTCOMES:
Oxygen desaturation index | Six months
Pulse rate | Six months
Endothelial dysfunction | Six months
Sleep quality and sleepiness | Six months
Health-related quality of life | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Kazuo Chin, MD, PhD, Principal Investigator — Graduate School of Medicine, Kyoto University; Toru Oga, MD, PhD, Principal Investigator — Graduate School of Medicine, Kyoto University
Locations (2):
- Japan (2):
  - Kirigaoka Tsuda Hospital, Kitakyushu
  - Kyoto University Hospital, Kyoto